CLINICAL TRIAL: NCT05900999
Title: Addressing Arm Non-use by Encouraging Idle-time Activity During Early Recovery From Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: Medical College of Wisconsin (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MCW PRO00042316 / MU HR-4044; 5R21HD106132-02 (NIH)
Record Dates: First submitted 2023-05-16; First posted 2023-06-13 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-10

CONDITIONS: Stroke; Exercise
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: Survivors of stroke in early stages of recovery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survivors of stroke in early stages of recovery (Experimental)
  Interventions: Behavioral: Feasibility of idle time exercise

INTERVENTIONS:
Behavioral: Feasibility of idle time exercise — The experiments in this proposal will assess the utility and subjective patient experience performing idle time exercise intervention designed to reduce learned non-use of the hemiparetic arm in the days, and weeks immediately following stroke. Exercise will be cued by wearable technology that provides vibrotactile cues similar to those provided by FitBit devices. Participants will be asked to perform simple exercises after receiving a vibration cue. In the first four sessions they will tap the more-involved wrist; in the second four sessions they will passively move the more-involved elbow through a range of motion; in the final four sessions they will actively move the more-involved elbow through a range of motion. Accelerometers in the wearable devices will monitor motion of the wrist during the exercise sessions. We will interview the participants two months later regarding how well they use the more-involved arm to perform daily activities.

SUMMARY:
This project evaluates the feasibility of using custom wearable technology and associated procedures to increase activity of the more-involved upper extremity during the earliest stages of recovery from stroke by increasing the amount of therapeutic exercise during idle-time. The proposed research is relevant to public health because it takes steps to mitigate a significant problem in physical rehabilitation using low-cost technology to motivate and monitor idle-time exercise without adding significantly to clinician workloads. The project aligns with the NICHD / NCMRR Research Plan on Rehabilitation by exploiting a mobile health (mHealth) and sensor-based approach to promote health and wellness through participant-engaged, data-driven, individualized care.

DETAILED DESCRIPTION:
The experiments in this proposal will assess the functional utility and subjective patient experience using a personal exercise cueing system designed to reduce learned non-use of the hemiparetic arm in the days, and weeks immediately following stroke. Up to 36 stroke survivors will be asked to participate in 12 practice sessions each lasting approximately 90 minutes. Participants will be asked to perform simple exercises after receiving a vibration cue. In the first four sessions participants will tap the more-involved wrist; in the second four sessions they will passively move the more-involved elbow through a range of motion; in the final four sessions they will actively move the more-involved elbow through a range of motion.

Accelerometers in the wearable devices will monitor motion of the wrist during the exercise sessions. To verify functional utility of the system, the investigators will examine for differences in the duration of arm movement activity in the cued exercise sessions relative to uncued periods. After all the sessions are complete, subjective user experience will be assessed by asking participants to complete a series of surveys wherein they can provide information about their subjective experiences with the wearable device technology. To assess feasibility of long-term follow-up, the investigators will interview the participants two months later regarding how well they use the more-involved arm to perform daily activities. At this time, they will also be asked to wear the devices for two days to assess the ability to measure arm movement activity at follow-up.

ELIGIBILITY:
Inclusion Criteria (General): The goal of this feasibility clinical trial is to assess the functional utility and subjective patient experience using a personal exercise cueing system designed to reduce learned non-use of the hemiparetic arm in the days, and weeks immediately following stroke. We therefore restrict inclusion to stroke survivors in the inpatient rehabilitation unit of Froedtert Memorial Hospital (Milwaukee, WI). Thus, candidate subjects will undergo screening by Dr. McGuire and his team prior to inclusion in the study. Stroke survivors shall have:

* had a unilateral stroke within the last 30 days;
* ability to give informed consent and be able to follow two-stage instructions;
* a broad range of motor impairment as assessed using the upper extremity portion of the Fugl-Meyer Motor Assessment (i.e., UE-FM score <= 50 out of a possible 66);
* age ≥ 18 yr. of age.

Exclusion Criteria (General) include:

* Inability of subjects to give informed consent or follow two-stage instructions;
* concurrent illness or severe pain limiting the capacity to conform to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Memorial Hospital, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data have been shared, as described in our recent manuscript (Bassindate et al., 2025: https://www.mdpi.com/2076-3417/15/6/3010).
Supporting Information: Analytic Code
Time Frame: * https://doi.org/10.5281/zenodo.14990338 (4 March 2025 onward; no end date).
  * https://www.mdpi.com/2076-3417/15/6/3010 (select Download -> Download Supplementary Material)
Access Criteria: Anyone with access to the web-links can access the data and analysis codes.

REFERENCES:
- [Result] Bassindale K, Golus S, Horder J, Winkoski M, Sytsma M, Morelli WA, Casadio M, McGuire J, Scheidt RA. The Feasibility and User Experience of a Program of Progressive Cued Activity to Promote Functional Upper Limb Activity in the Inpatient Rehabilitation Setting with Follow-Up at Home. Appl Sci (Basel). 2025 Mar 2;15(6):3010. doi: 10.3390/app15063010. Epub 2025 Mar 11. PMID 40727538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: 11/29/2022 through 7/18/2023. Recruitment location: inpatient rehabilitation facility
Groups:
- Survivors of Stroke in Early Stages of Recovery: This was a single cohort study. We evaluated the feasibility, functional utility, and subjective user experience of a progressive-challenge cued activity program, delivered via wearable technology, to promote upper limb activity in an inpatient rehabilitation facility during the early days and weeks following stroke.
  Quantitative movement data was collected using accelerometry (motion trackers worn on both wrists) to estimate compliance with the cue responses. We assessed user experience using validated quantitative surveys that measure motivation to engage with the system, perceptions of system usability, and the degree of user satisfaction while using the technology.
Period: Overall Study
Arm/Group | Survivors of Stroke in Early Stages of Recovery
Started | 42
Completed | 30
Not Completed | 12
Not completed — Withdrawal by Subject | 9
Not completed — transfer to another facility; too complex of a therapy schedule; physician withdrawal | 3

BASELINE CHARACTERISTICS:
Population: Of the 42 recruited participants, 12 withdrew or were withdrawn. Reasons for withdrawal included: disliking the vibrotactile cues after initial demonstration with the device (4), disliking the cues after 1-2 days of use (5), transfer of care to outside facility (1), complex therapy schedule (1), and physician withdraw (1).
Arm/Group | Survivors of Stroke in Early Stages of Recovery
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] — units of measure: years
  Years | 63.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: numerical score (ordinal)] — a screening tool to assess cognitive ability (max score: 30; scores 26 to 30 indicate normal cognition; scores 18-25 indicate mild cognitive impairment; scores 10-19 indicate moderate impairment; scores 0-9 indicate severe impairment) Population: 12 participants withdrew or were withdrawn
  numerical score (ordinal)
    number analyzed (Participants) | 30
    (all) | 25.9 (4.2)
Fugl-Meyer Upper Extremity Motor Score [Mean (Standard Deviation); unit: numerical score (ordinal)] — Possible score range: 0 (most impaired) to 66 (unimpaired)
  numerical score (ordinal) | 45.6 (25.1)
Fugl-Meyer Upper Extremity Sensory Score [Mean (Standard Deviation); unit: numerical score (ordinal)] — Possible score range: 0 (most impaired) to 12 (unimpaired)
  numerical score (ordinal) | 11.5 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Average Activity Duration (RAAD)
Description: The RAAD assesses the amount of measured arm activity during cued exercise epochs compared to non-cued epochs. A RAAD value greater than 1.0 indicates that the amount of arm activity in response to Souvenir cues exceeded the amount of activity during non-cued periods of time.
Time Frame: During device use in an inpatient setting (about 1 to 3 weeks of use).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Survivors of Stroke in Early Stages of Recovery
Number analyzed (Participants) | 30
ratio | 1.223 (0.63)

2. Primary Outcome: System Usability Scale
Description: The System Usability Scale (SUS) assesses the usability of the activity cueing system and monitoring system within the context of encouraging therapeutic arm activity. Scores are provided on a scale ranging from 1 to 100, with higher scores indicating greater perceived usability. Scores greater than 68 are generally considered to indicate "passable" usability.
Time Frame: Two time points: After device use in an inpatient setting (after about 1 to 3 weeks of use); after device use in home settings (after 2 days of use).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Survivors of Stroke in Early Stages of Recovery
Number analyzed (Participants) | 30
units on a scale
  SUS obtained after using the device in an inpatient setting | 80.1 (13.8)
  SUS obtained after using the device in home settings: number analyzed (Participants) | 23
  SUS obtained after using the device in home settings | 83.3 (15.2)

3. Primary Outcome: Intrinsic Motivation Inventory (IMI)
Description: The IMI assesses subjective experience of motivation in response to the system's vibrotactile cues. IMI comprises 37 questions, with answers provided on a Likert scale (1-7).
  IMI questions span 6 psychosocial dimensions:
  * interest/enjoyment; higher scores = more interest/enjoyment with cued activities
  * effort/importance; higher scores = more perceived importance and more effort put into performing cued activities
  * value/usefulness higher scores = more perceived value and usefulness of cued activities
  * perceived choice; higher scores = greater degree to which participants felt that they had choice in engaging with the cued activities
  * perceived competence; higher scores = greater degree of competence performing cued activities
  * pressure/tension; higher scores = more anxiety/tension performing cued activities.
  A composite score is computed within each dimension by averaging item responses after reversing specified negative items; a score of 4 separates (+) from (-) experiences.
Time Frame: After device use in an inpatient setting (after about 1 to 3 weeks of use).
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Survivors of Stroke in Early Stages of Recovery
Number analyzed (Participants) | 30
units on a scale
  interest/enjoyment dimension | 4.9 (1.3)
  effort/importance dimension | 5.4 (1.4)
  value/usefulness dimension | 6.2 (0.9)
  perceived choice dimension | 6.0 (0.9)
  perceived competence dimension | 5.8 (1.2)
  pressure/tension dimension | 2.8 (1.0)

4. Primary Outcome: Quebec User Evaluation of Satisfaction With Technology (QUEST)
Description: The QUEST assesses user satisfaction with the system and its delivery by the research team.. The QUEST comprises 12 questions, with answers provided on a Likert scale (1-5). For each question, a score of "1" = not at all satisfied where "5" is "very satisfied". A composite score (min = 1; max = 5) is computed for the QUEST by averaging across all questions. A score of 3 separates (+) from (-) experiences.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Survivors of Stroke in Early Stages of Recovery
Number analyzed (Participants) | 30
units on a scale
  QUEST post-device use in an inpatient setting | 4.52 (0.46)
  QUEST after use in home settings: number analyzed (Participants) | 23
  QUEST after use in home settings | 4.5 (0.5)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up (up to 6 months post-discharge)
Arm/Group | Survivors of Stroke in Early Stages of Recovery
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT05900999/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT05900999/ICF_001.pdf